CLINICAL TRIAL: NCT04734470
Title: Expression of CD19 Complex in Lymphoproliferative Disorders
Acronym: CD19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahran mohamed hussein mahran, Doctor, Assiut University
Other Study IDs: Expression of CD19 complex
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Lymphoproliferative Disorders
MeSH Terms: conditions — Lymphoproliferative Disorders | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Flow cytometry — The study of CD19 complex expression in lymphoproliferative disorders by flowcytometry

SUMMARY:
1. To study the expression pattern of CD19(cluster of differentiation antigen19) complex in lymphoproliferative disorders and its diagnostic value.
2. To investigate the biological significance of CD19 complex expression in lymphoproliferative disorders.
3. To explore the possibility of ectopic expression of CD19 complex in non B-lineage lymphoproliferative disorders.

DETAILED DESCRIPTION:
Lymphoproliferative disorders (LPD)comprise a heterogeneous group of diseases characterized by uncontrolled production of lymphocytes that cause monoclonal lymphocytosis, lymphadenopathy and bone marrow infiltration.They Typically occur in people who have a compromised immune system with highly variable clinical course.

Lymphoproliferative disorders are immunomorphologically and clinically heterogeneous. The two major types of lymphocytes are B cells and T cells, which are derived from pluripotent hematopoietic stem cells in the bone marrow.

Lymphoproliferative disorders include; Follicular lymphoma, chronic lymphocytic leukemia, acute lymphoblastic leukemia, hairy cell leukemia, Hemophagocytic lymphohistiocytosis (HLH), B-cell lymphomas, T-cell lymphomas, multiple myeloma, Waldenström's macroglobulinemia, Wiskott Aldrich syndrome, Langerhans cell histiocytosis (LCH), Lymphocyte-variant hypereosinophilia, Pityriasis Lichenoides, post-transplant lymphoproliferative disorder, autoimmune lymphoproliferative syndrome (ALPS), Lymphoid interstitial pneumonia, Epstein Barr virus associated lymphoproliferative diseases, Castleman disease and X-linked lymphoproliferative disease.

Many patients are asymptomatic at the time of first presentation, with the diagnosis being made as an incidental finding after a routine medical examination or blood test, for example, complete blood count (CBC).

Definitive diagnosis is made on the characteristic lymphocyte morphology and immunophenotype usually from samples of peripheral blood ,bone marrow samples or lymph nodes.

The membrane receptor proteins (CD19, CD81, CD21 (complement receptor type2) and Leu-13(CD225)), form a complex (CD19 complex) on human B lymphocytes that has costimulatory activity for the antigen receptor, membrane IgM(mIgM) .The complex is unique among known membrane protein complexes of the immune system because its components represent different protein families, and can be expressed individually.

The biochemical mechanism by which the complex costimulates is not understood.CD19 has been shown to be a major substrate of a protein tyrosine kinase activated by mIgM, and tyrosine phosphorylated CD19 binds phosphatidylinositol 3-kinase (PI3-kinase), an enzyme that is required for the cellular activating effects of certain receptor tyrosine kinases. Thus, several biochemical pathways may be triggered by the CD21/CD19/CD81/CD225 complex that relate to its role in amplifying the response of B cells to antigen.

Multiple biologic effects of the CD21/CD19/ CD81/CD225 complex may reflect the discrete actions of individual components, each of which is a member of a distinct protein family: CD21 of the regulators of complement activation family; CD19 of the Ig superfamily;and CD81 of the tetraspan family of membrane proteins and is an important regulator of B-cell signaling. CD225 of Interferon-induced transmembrane protein (IFITM) family.

Although CD19 function may be elicited following its potential binding to an as yet unidentified ligand, C3d binding to CD21 supplies an already characterized ligand for the CD19 complex, thereby linking complement immune responses and the generation of immunological activation and B cell function.

Ligation of members of the CD19 complex initiates a cascade of biological responses that can modulate signal transduction through the B cell Ag-receptor complex and other cell surface receptors. So it may help in understanding the signal transduction pathways through this complex.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute lymphoproliferative disorders.
* Patients with chronic lymphoproliferative disorders

Exclusion Criteria:

* patients with non lymphoid disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sample size is 92 (46 in each arm) but number of controls will be decreased and number of cases will be increased.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
To study the expression pattern of CD19 complex in lymphoproliferative disorders and its diagnostic value. | Baseline
  Study of CD19 complex expression pattern in lymphoproliferative disorders by flow cytometry

REFERENCES:
- [Background] Goede V, Fischer K, Busch R, Engelke A, Eichhorst B, Wendtner CM, Chagorova T, de la Serna J, Dilhuydy MS, Illmer T, Opat S, Owen CJ, Samoylova O, Kreuzer KA, Stilgenbauer S, Dohner H, Langerak AW, Ritgen M, Kneba M, Asikanius E, Humphrey K, Wenger M, Hallek M. Obinutuzumab plus chlorambucil in patients with CLL and coexisting conditions. N Engl J Med. 2014 Mar 20;370(12):1101-10. doi: 10.1056/NEJMoa1313984. Epub 2014 Jan 8. PMID 24401022
- [Background] Zavala-Vega S, Palma-Lara I, Ortega-Soto E, Trejo-Solis C, de Arellano IT, Ucharima-Corona LE, Garcia-Chacon G, Ochoa SA, Xicohtencatl-Cortes J, Cruz-Cordova A, Luna-Pineda VM, Jimenez-Hernandez E, Vazquez-Meraz E, Mejia-Arangure JM, Guzman-Bucio S, Rembao-Bojorquez D, Sanchez-Gomez C, Salazar-Garcia M, Arellano-Galindo J. Role of Epstein-Barr Virus in Glioblastoma. Crit Rev Oncog. 2019;24(4):307-338. doi: 10.1615/CritRevOncog.2019032655. PMID 32421988
- [Background] Vaillant AAJ, Stang CM. Lymphoproliferative Disorders. StatPearls [Internet]: StatPearls Publishing; 2020.
- [Background] Zheng YY, Chen G, Zhou XG, Jin Y, Xie JL, Zhang SH, Zhang YN. [Retrospective analysis of 4 cases of the so-called blastic NK-cell lymphoma, with reference to the 2008 WHO classification of tumours of haematopoietic and lymphoid tissues]. Zhonghua Bing Li Xue Za Zhi. 2010 Sep;39(9):600-5. Chinese. PMID 21092587
- [Background] Byrd JC, Brown JR, O'Brien S, Barrientos JC, Kay NE, Reddy NM, Coutre S, Tam CS, Mulligan SP, Jaeger U, Devereux S, Barr PM, Furman RR, Kipps TJ, Cymbalista F, Pocock C, Thornton P, Caligaris-Cappio F, Robak T, Delgado J, Schuster SJ, Montillo M, Schuh A, de Vos S, Gill D, Bloor A, Dearden C, Moreno C, Jones JJ, Chu AD, Fardis M, McGreivy J, Clow F, James DF, Hillmen P; RESONATE Investigators. Ibrutinib versus ofatumumab in previously treated chronic lymphoid leukemia. N Engl J Med. 2014 Jul 17;371(3):213-23. doi: 10.1056/NEJMoa1400376. Epub 2014 May 31. PMID 24881631
- [Background] van Zelm MC, Reisli I. CD19 Deficiency due to Genetic Defects in the CD19 and CD81 Genes. Humoral Primary Immunodeficiencies: Springer; 2019. p. 83-95.
- [Background] Pongas GN, Annunziata CM, Staudt LM. PI3Kdelta inhibition causes feedback activation of PI3Kalpha in the ABC subtype of diffuse large B-cell lymphoma. Oncotarget. 2017 Sep 13;8(47):81794-81802. doi: 10.18632/oncotarget.20864. eCollection 2017 Oct 10. PMID 29137222
- [Background] Dasgupta S, Dasgupta S, Bandyopadhyay M. Regulatory B cells in infection, inflammation, and autoimmunity. Cell Immunol. 2020 Jun;352:104076. doi: 10.1016/j.cellimm.2020.104076. Epub 2020 Feb 27. PMID 32143836
- [Background] Feingold JM, Ungar DR. DOSAGE REGIMES FOR THE ADMINISTRATION OF AN ANTI-CD19 ADC. US Patent App. 16/622,649; 2020.
- [Background] Beckwith KA, Byrd JC, Muthusamy N. Tetraspanins as therapeutic targets in hematological malignancy: a concise review. Front Physiol. 2015 Mar 23;6:91. doi: 10.3389/fphys.2015.00091. eCollection 2015. PMID 25852576
- [Background] Yanez DC, Ross S, Crompton T. The IFITM protein family in adaptive immunity. Immunology. 2020 Apr;159(4):365-372. doi: 10.1111/imm.13163. Epub 2019 Dec 22. PMID 31792954
- [Background] Carroll MC. The complement system in B cell regulation. Mol Immunol. 2004 Jun;41(2-3):141-6. doi: 10.1016/j.molimm.2004.03.017. PMID 15159059
- [Background] Tedder TF, Poe JC, Fujimoto M, Haas KM, Sato S. The CD19-CD21 signal transduction complex of B lymphocytes regulates the balance between health and autoimmune disease: systemic sclerosis as a model system. Curr Dir Autoimmun. 2005;8:55-90. doi: 10.1159/000082087. PMID 15564717